CLINICAL TRIAL: NCT06486532
Title: HeartBeet Clinic Randomized Pilot Trial
Brief Title: HeartBeet Clinic Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Principal Investigator, Stephanie Hooker, Research Investigator, HealthPartners Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A24-048
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-06

CONDITIONS: Hyperlipidemia; Hypertension
Keywords: Cardiovascular health
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HeartBeet Clinic (Experimental): 16 week group based lifestyle intervention
  Interventions: Behavioral: HeartBeet Clinic
- Self-paced education (Active Comparator): Online learning of lifestyle medicine
  Interventions: Behavioral: Self-paced education

INTERVENTIONS:
Behavioral: HeartBeet Clinic — 16 weeks of group based lifestyle medicine coaching covering the six pillars of lifestyle medicine. The six pillars of lifestyle medicine include regular physical activity; a whole-food plant-based diet; restorative sleep; limiting substance use (e.g., tobacco and alcohol use); having meaningful social connections; and stress management. Groups will be led by clinician or health coach expert.
  Arms: HeartBeet Clinic
Behavioral: Self-paced education — Self-paced course and workbook with no contact with study clinician or health coach expert
  Arms: Self-paced education

SUMMARY:
The goal of the current study is to conduct a pilot randomized controlled trial comparing the HeartBeet Clinic, a 16-week lifestyle medicine program with virtual, small-group coaching, to a self-paced, online education program. In this pilot study, the primary goals will be to assess acceptability and feasibility of the study and intervention procedures to prepare for a larger efficacy trial.

DETAILED DESCRIPTION:
Individuals randomized to the 16-week HeartBeet Clinic lifestyle medicine intervention will complete two in-person group visits, one at the beginning and one at the end of the program. They will also attend group coaching sessions that will be held virtually, using an online coaching platform that will house the self-paced course, intervention materials, and schedule for the coaching and live events. Individuals in this group will be asked to attend 12 group coaching sessions with a health coach, 6 skills sessions to enhance behavior change skills with a health coach, and 6 deep dives with subject matter experts. These sessions will require 1-2 hours of participation per week. In addition, participants will be asked to work through the self-paced course and workbook activities on their own between sessions.

Individuals randomized to the self-paced education group will have access to the virtual coaching platform for the self-paced course and workbook. They will receive email reminders to work through the workbook activities. They will not have contact with the study clinician or health coach except to troubleshoot technical issues.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one cardiovascular risk factor, including: a) high cholesterol, as defined as diagnosis of hyperlipidemia and/or most recent total cholesterol > 200 or b) hypertension (as defined by a diagnosis of hypertension and/or active antihypertensive medication prescription) and/or BMI > 27
* Identify as a HealthPartners patient, including having an outpatient encounter with a HealthPartners or Park Nicollet clinician in the prior year
* Be willing to pay for copays/charges for group medical visit and labs drawn as part of usual care if not fully covered by insurance
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Willingness to maintain current doses of statin, anti-obesity medication, and/or antihypertensive medication during the study
* Willingness and ability to attend weekly group coaching sessions for 16 weeks at ≥ 1 scheduled group coaching time
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access

Exclusion Criteria:

* Concurrent participation in another treatment or intervention study
* History of coronary artery, cerebrovascular or peripheral arterial disease including myocardial infarction, unstable angina, revascularization, stroke/TIA, carotid intervention, claudication, or congestive heart failure
* Existing diagnosis of dementia and/or other cognitive impairment that would be a barrier to participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Acceptability | Within 2 weeks post-intervention
  Assess the acceptability using Client Satisfaction Questionnaire (CSQ-8; Larsen et al., 1979). Participants report the extent to which the intervention met their expectations on a 8-item scale. Participants rate the quality of the service and their satisfaction with the services provided on a 4-point Likert-type scale with varying response options (e.g., "How would you rate the quality of the service you received? 4 = Excellent, 3 = Good, 2 = Fair, or 1 = Poor). Items were summed for a total score ranging from 8 to 32, with higher scores corresponding to greater satisfaction with treatment.

SECONDARY OUTCOMES:
Recruitment and Retention feasibility | End of study (5 months)
  Assess feasibility of the intervention based on meeting recruitment and retention targets.
Cardiovascular health | Within 2 weeks post-intervention
  Cardiovascular health will be measured by Life's Essential 8 (Lloyd-Jones et al., 2022), a composite measure that includes 8 domains: diet quality, physical activity, smoking, sleep, lipids, blood pressure, blood glucose, and body mass index. Each domain is scored on a scale from 0-100; a total cardiovascular health score is the average of the 8 domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Park Nicollet Cardiology, Saint Louis Park, Minnesota, United States